CLINICAL TRIAL: NCT05103137
Title: Post-transition Clinical and Socio-professional Future in Adult Patients With Recurrent Multifocal Chronic Osteitis
Acronym: ESPERANTO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0481
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Chronic Recurrent Multifocal Osteomyelitis
MeSH Terms: conditions — Chronic recurrent multifocal osteomyelitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaires concerning assesment of quality of life with 3 different questionnaires ( SF36, HAQ and pre-established questionnaire for the study) during a phone interview

SUMMARY:
Chronic Recurrent Multifocal Osteomyelitis (CRMO) is a rare autoinflammatory bone disease in children. Studies evaluating the quality of life of patients with CRMO are small and heterogeneous. A better understanding of the impact of the disease on the quality of life of adult patients with CRMO beginning in childhood would allow better long-term management of these patients. Our study aims are to assess the clinical and socio-professional outcomes of adult patients who started CRMO at pediatric age.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient with a CRMO with pediatric-onset disease (> 18years)
* Patient who was informed and agreed to participate in this study

Exclusion Criteria:

* Patients with Monogenic auto-inflammatory disease associated with osteolytic bone lesions (e.g. interleukin-1 receptor antagonist deficiency)
* Patient with Majeed syndrome
* Patient without sufficient imaging data to confirm the presence of one or more inflammatory lesions
* Patients with incomplete data.
* Patients placed under legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CRMO disease started at pediatric age. Patients who agreed to participate to the study (study questionnaires during a telephone interview (SF36, HAQ and questionnaire pre-established for the study)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Impact of the disease on the quality of life of adult CRMO patients with pediatric-onset disease. | 20 minutes
  Result of the SF 36 (Short Form 36) quality of life questionnaire compared to data in the general population and other published data available in CRMO and inflammatory diseases in children.
  This questionnaire is composed of 36 questions which allow to calculate two scores of the quality of life of individuals: the physical composite score (SCP) and the mental composite score (SCM). The higher the score the higher the capacity.
  Range 0 to 100

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service Rhumatologie Pédiatrique Centre De Référence Maladies Rares RAISE Hôpital Femme Mère Enfant, Bron
  - Service de Rhumatologie Centre Hospitalier Edouard Herriot, Lyon
  - Service de Rhumatologie Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No